CLINICAL TRIAL: NCT04047589
Title: Assessing Exercise Behavior and Preferences Among Patients and Oncologists at Indiana University Simon Cancer Center
Brief Title: Assessing Exercise Behavior and Preferences Among Patients and Oncologists
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tarah J Ballinger, MD, Assistant Professor of Clinical Medicine, Indiana University
Other Study IDs: IUSCC-0690
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumor; Exercise
Keywords: solid tumor; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects: Cancer patients with curable or previously treated malignancies
  Interventions: Behavioral: Survey regarding exercise habits, barriers to exercise, and experience with exercise services from the cancer center.
- Providers: Physicians seeing patients in the outpatient clinics at the IU Simon Cancer Center
  Interventions: Behavioral: Survey regarding personal exercise habits and beliefs, barriers to making exercise recommendations

INTERVENTIONS:
Behavioral: Survey regarding exercise habits, barriers to exercise, and experience with exercise services from the cancer center. — Survey created at Indiana University to gain information regarding exercise habits, barriers to exercise, and experience with exercise services from the cancer center.
  Groups: Subjects
Behavioral: Survey regarding personal exercise habits and beliefs, barriers to making exercise recommendations — Survey regarding personal exercise habits and beliefs, barriers to making exercise recommendations, and potential resources the cancer center might provide to help make effective exercise recommendations in the future
  Groups: Providers

SUMMARY:
The purpose of this study is to understand the preferences and barriers surrounding exercise of both the patients and oncologists within Indiana University Simon Cancer Center. This information will establish gaps in our current care and provide important information to guide future pilot interventions.

DETAILED DESCRIPTION:
This descriptive, cross-sectional study will survey patients with a current or previous diagnosis of non-metastatic solid tumor malignancy who are being seen at the Indiana University Simon Cancer in Indianapolis, Indiana. Patients with active, incurable disease are excluded. Willing and eligible patients will complete a brief, 14 question survey while seen in the waiting room of the women's or multi-disciplinary clinics. We aim to survey 350 patients over a 12 month period. Patients will fill out the survey at only one point in time and no patient identifiers will be kept.

During COVID-19 restrictions, we will also send out an electronic version of the survey to participants using the email address provided in their Cerner accounts. Responses will be captured by REDCAP and will remain anonymous and not linked to the patients' medical record or personal health information.

The physician survey will be emailed to oncologist/hematologists practicing within IUSCC who see patients at least once per week. Physicians will receive a survey at only one point in time. The survey will be anonymous and no physician identifiers will be kept.

Primary objective Estimate the proportion of patients with curable solid tumor malignancies seen at the Indiana University Simon Cancer Center who are meeting exercise recommendations for cancer survivors (more than 150 minutes per week of moderate or 75 minutes per week of vigorous activity).

Secondary objectives

* Assess patients' perceived barriers to exercise during cancer survivorship
* Assess patients' preferences for receiving exercise recommendations
* Assess oncologists' perceived barriers to making exercise recommendations
* Assess oncologists' preferences for exercise and physical activity resources that could be provided by the cancer center

ELIGIBILITY:
Inclusion Criteria:

* Physician survey Any oncologist/hematologist practicing within IUSCC regularly providing care for patients with solid tumor malignancies (seeing patients one or more days per week in the multidisciplinary or women's clinics with solid tumor malignancies). Physicians providing care only for hematologic (multiple myeloma, leukemia, lymphoma, transplant) or benign disorders will be excluded.
* Patient survey

  1. Patients with a current or previous diagnosis of stage 0-III or curable solid tumor
  2. Patients receiving any component of their medical oncologic care at IUSCC
  3. Age ≥ 18 years
  4. Able to read and write English

Exclusion Criteria:

1. Metastatic disease at the time of study participation
2. Inability to complete the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential patients will be identified in the outpatient clinics (women's and multi-disciplinary) at the IU Simon Cancer Center. Physicians will be given the option of requesting that their patients not participate in the survey. When patients check in or are placed in an exam room, a trained member of the clinic staff will approach patients about possible participation in the survey study.
  Physicians seeing patients more than once per week in the outpatient clinics at the IU Simon Cancer Center will receive email invitation to participate in the survey. An online survey will be administered via Survey Monkey. This does not require an informed consent process. The survey has 14 questions and will take approximately 5 minutes to complete.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who meet exercise recommendations. | baseline
  Patients self-reporting more than 150 minutes per week of moderate physical activity OR more than 75 minutes per week of vigorous physical activity

SECONDARY OUTCOMES:
Patient Perceived barriers to exercise during cancer survivorship via pilot survey | Baseline
  Investigator created survey with 14 items regarding demographics, cancer history, exercise habits, and exercise as part of cancer treatment
Patient preferences for receiving exercise recommendations via pilot survey | Baseline
  Investigator created survey with 14 items regarding demographics, cancer history, exercise habits, and exercise as part of cancer treatment
Provider perceived barriers to making exercise recommendations via pilot survey | Baseline
  Investigator created survey with 14 items regarding demographics, cancer speciality, exercise habits, and exercise recommendations to patients and patient exercise habits
Provider preferences for exercise and physical activity resources that could be provided by the cancer center via pilot survey | Baseline
  Investigator created survey with 14 items regarding demographics, cancer speciality, exercise habits, and exercise recommendations to patients and patient exercise habits

CONTACTS AND LOCATIONS:
Overall Officials: Tarah Ballinger, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana, United States